CLINICAL TRIAL: NCT00391781
Title: Prospective Randomised Controlled Trian of Warmed vs. Room Temperature Contrast Media for Hystersalpingography
Brief Title: Warm Contrast Media for Pain Reduction During Hystersalpingography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: WARMHSG.CTIL
Record Dates: First submitted 2006-10-23; First posted 2006-10-24 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-08

CONDITIONS: Infertility
Keywords: mechanical infertility; hysterosalpingogram; hysterosalpingography
MeSH Terms: conditions — Infertility

INTERVENTIONS:
Procedure: Temperature of contrast medium

SUMMARY:
The aim of this study is to compare between body-temperature to room-temperature contrast media used during hysterosalpingography. We hypothesize that warmed medium will reduce pain associated with the procedure.

DETAILED DESCRIPTION:
Infertility occurs in about 15% of all couples. One of the common methods for evaluation of mechanical infertility is hysterosalpingography (HSG). Several reports have shown that this common procedure is associated with moderate pain, i.e. around 5 on a visual analog scale (VAS)of 1-10. It is therefore important to find modes for pain reduction for HSG. According to a report on sonohydrosonograpy, a similar technique using sonography, insertion of media warmed to body temperature into the uterus significantly reduced the pain during the procedure compared with media at room-temprature. The use of room-temperature media is the routine in our institution, as well as in many others. A comparison between the media at different temperatures has not been reported so far.

We plan to perform a prospective trial in which patients referred for HSG will be randomized to the procedure using either warmed or room-temperature media. we will asses pain levels using VAS during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: infertility
* sex: female
* age: 18-45

Exclusion Criteria:

* active pelvic inflammotory disease
* known sensitivity to contrast medium

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2006-12; Study Completion 2008-12

PRIMARY OUTCOMES:
Pain level

CONTACTS AND LOCATIONS:
Overall Officials: Avi Tsafrir, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- women's health center, Ramot Eshkol, Jerusalem, Israel

REFERENCES:
- [Background] Nirmal D, Griffiths AN, Jose G, Evans J. Warming Echovist contrast medium for hysterocontrastsonography and the effect on the incidence of pelvic pain. A randomized controlled study. Hum Reprod. 2006 Apr;21(4):1052-4. doi: 10.1093/humrep/dei440. Epub 2005 Dec 22. PMID 16373408